

| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| Туре | Version | Document Identifier | Effective Date |
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


#### **CONFIDENTIAL**

#### STATISTICAL ANALYSIS PLAN FOR PROTOCOL 207640

Determination of the Sun Protection Factor of a Cosmetic Daily Defence Skin Cream

# BIOSTATISTICS DEPARTMENT GLAXOSMITHKLINE CONSUMER HEALTHCARE

Document type: Statistical Analysis Plan

Authors: PPD (Statistician II)

Document status: Final 1.0

Release date: 29-Jun-2017

Property of GSK Consumer Healthcare
May not be used, divulged, published or otherwise disclosed
without the consent of GSK



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

# **Table of contents**

| | Table | of conter | nts | 2 |
|---|---|---|---|---|
| 1 | Study | details | | 4 |
| | 1.1 | Study d | esign | 4 |
| | 1.2 | Study o | bjectives | 6 |
| | 1.3 | Treatme | ents | 7 |
| | 1.4 | Timepo | vints and visit windows | 7 |
| 2 | Data a | analysis | | 7 |
| | 2.1 | Populat | ions for analysis | 7 |
| | | 2.1.1 | Subject disposition | 7 |
| | | 2.1.2 | Protocol violations | 8 |
| | | 2.1.3 | Analysis populations | 8 |
| | | 2.1.4 | Subgroups/Stratifications | 8 |
| | | 2.1.5 | Centers pools | 8 |
| | 2.2 | Patient | demographics/other baseline characteristics | 8 |
| | | 2.2.1 | Demographic characteristics | 9 |
| | | 2.2.2 | General medical history | 9 |
| | | 2.2.3 | Characteristics of Disease | 9 |
| | 2.3 | | ents (study drug, rescue medication, other concomitant therapies, ance) | 10 |
| | | 2.3.1 | Study Product/drug Compliance and Exposure | 10 |
| | | 2.3.2 | Concomitant medication | 10 |
| | 2.4 | Analysi | s of Sun Protection Factor (SPF) | 10 |
| | | 2.4.1 | Primary efficacy endpoint | 10 |
| | | 2.4.2 | Secondary efficacy endpoint | 11 |
| | | 2.4.3 | Handling of missing values/censoring/discontinuations | 11 |
| | 2.5 | Analysi | s of secondary objectives | 11 |
| | 2.6 | Safety. | | 11 |
| | 2.7 | Analysi | s of other variables | 11 |
| | 2.8 | Interim | analysis | 12 |
| | 2.9 | Sample | size calculation | 12 |
| 3 | Chang | ges to the | Protocol Defined Statistical Analysis Plan | 12 |
| 4 | Apper | ndix 1: | | 13 |
| | 4.1 | List of | Tables, Listings and Figures | 13 |
| | 4.2 | Tables. | | 13 |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

| | 4.3 | Listings | 13 |
|---|-------|------------------------------------------------|----|
| | 4.4 | Top line Outputs | 14 |
| 5 | Appei | ndix 2: | 15 |
| | 5.1 | Templates for the Tables, Listings and Figures | 15 |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

The purpose of this Statistical Analysis Plan (SAP) is to describe the planned analyses and output to be included in the Clinical Study Report for Clinical Study Protocol (CSP) 207640. This SAP will be finalized prior to database freeze and treatment code un-blinding.

## 1 Study details

An important parameter of efficacy for sunscreen products is the Sun Protection Factor (SPF). The SPF is a measure of how much solar energy (UV radiation) is required to produce sunburn on protected skin (i.e. in the presence of sunscreen) relative to the amount of solar energy required to produce sunburn on unprotected skin. In this study, the SPF is to be determined according to the International Standards Organization (ISO) 24444:2010 methodology (In vivo determination of the sun protection factor).

General safety and tolerability will be assessed based on the frequency and severity of Adverse Events (AEs).

### 1.1 Study design

#### **Overall Design**

A single-center, randomized, evaluator blind, intra-individual comparison, no treatment and positive controlled clinical study to determine the SPF of Physiogel Daily Defence Protective Day Cream Light as per ISO 24444:2010.

The provisional minimal erythemal dose of unprotected skin (MEDu) for each subject will be determined before starting the main test in order to center the UV dose ranges for the exposures of MEDu and MEDp. As the first step, a virgin area of skin on the back will be exposed to a preliminary series of UV exposures. The location of the irradiated test site for the provisional MEDu measurement will be randomised for all subjects. In this study, there will be a total of four irradiated test sites. Two test sites will be located below the scapula line, either side of the spine. The remaining two areas will be located below these sites and above the waist.

Six exposure sub-sites positioned within the randomised test area and centered on the estimated MEDu will be exposed to incremental UV doses using a geometric progression of 1.25. The dose of UV radiation administered will be chosen so that the estimated MEDu will be irradiated at the 4th of the 6 sub-sites. The estimated MEDu will be predicted based on the subject's mean Individual Typology Angle (ITA°) value. As the second step, a trained evaluator will assess the irradiated sub-sites for signs of unambiguous erythema 16-24 hours after UV exposure to determine the provisional MEDu. The provisional MEDu will be the lowest dose of UV radiation that produces the first perceptible unambiguous erythema with defined borders appearing over most of the field of UV exposure.

Once the provisional MEDu for a subject has been determined, the three remaining test sites will be demarcated. The test product (Physiogel Daily Defence Protective Day Cream Light) and positive control (P3 reference sunscreen formulation) will be applied to two of the three virgin test sites. The other test site will remain unprotected. The order of product application



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

(test product, reference product and unprotected test site) will be randomised over the entire test group. Once the test product and positive control have been applied to the assigned test sites, the subject will undergo a second series of incremental UV exposures. For the unprotected site, the range of UV doses administered shall be selected using the subject's provisional MEDu. Six exposure sub-sites centered on the provisional MEDu shall be exposed with incremental UV doses using a geometric progression of 1.25. The dose of UV radiation administered to subjects will be chosen such that the provisional MEDu will be irradiated at the 4th of the 6 sub-sites. For the product protected sites, the UV doses administered shall be selected using the subject's expected MEDp, which is the multiple of the provisional MEDu for the subject and the expected SPF of either the test product (21) or reference sunscreen formulation (16). A minimum of 6 sub-sites centered on the expected MEDp shall be exposed with incremental UV doses using a geometric progression of 1.25. The dose of UV radiation administered to subjects will be chosen such that the expected MEDp will be irradiated at the 4th of the 6 subsites.

The minimum number of valid individual SPF (SPFi) results shall be 10 and the maximum number of valid SPFi results shall be 20. In order to achieve between 10 and 20 valid results, a maximum of five individual invalid results may be excluded from the calculation of the mean SPF. Consequently the actual number of test subjects used will fall between a minimum of 10 and a maximum of 25 subjects (i.e. a maximum of 20 valid results plus 5 rejected invalid results).

The study will include subjects of more than one Fitzpatrick phototype (I, II or III). It will not be permitted to adjust the expected SPF of the test product from subject to subject.

#### Visit 1 – Subject Screening

The following assessments will be conducted:

- 1. Informed Consent
- 2. Demographics
- 3. Medical History
- 4. Current / Concomitant Medication
- 5. ITA° Measurement
- 6. Fitzpatrick Skin Type Assessment
- 7. In/Exclusion Criteria
- 8. Subject Eligibility

#### Visit 2 – Provisional MED Irradiation (UV Exposure)

The following assessments will be conducted:

- 1. Current / Concomitant Medication\*
- 2. Continued Eligibility\*
- 3. Exclusion Criteria\*
- 4. Subject Eligibility\*
- 5. Randomisation
- 6. Provisional Minimum Erythemal Dose (MED) Irradiation
- 7. Adverse Events
- \*Not required if Visit 2 is combined with Visit 1



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

#### Visit 3 – Provisional MED Evaluation

The following assessments will be conducted:

- 1. Current / Concomitant Medication
- 2. Continued Eligibility
- 3. Visual Grading of Exposure Sub-Sites (Test Sites)\*
- 4. Adverse Events
- \*Visual grading of skin must occur 16-24 hours after completion of the Provisional MED Irradiation procedure

#### **Visit 4 – Test Irradiation (UV Exposure)**

The following assessments will be conducted:

- 1. Current / Concomitant Medication\*
- 2. Continued Eligibility\*
- 3. Test Product and Reference Sunscreen Application to Randomly Assigned Test Sites on the Back
- 4. UV Exposure of Test Product Treated, Reference Sunscreen Formulation Treated and Unprotected Test Sites
- 5. Adverse Events
- \*Not required if Visit 4 is combined with Visit 3

# Visit 5 – MEDp and MEDu Determination and SPF Calculation for Test and Reference Sunscreen

The following assessments will be conducted:

- 1. Current / Concomitant Medication
- 2. Continued Eligibility
- 3. Visual Grading of Exposure Sub-Sites to Determine MEDp and MEDu and calculate SPF\*
- 4. Adverse Events
- 5. Subject Discharge from Study
- \* Visual grading of skin must occur 16-24 hours after completion of the Test Irradiation procedure

## 1.2 Study objectives

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To determine the Sun Protection Factor of the test product | Arithmetic mean of all valid individual sun protection factor (SPFi) values; where SPFi = Minimal Erythemal Dose of product treated (MEDp) test sites in relation to unprotected (MEDu) test sites 16-24 hours after exposure to ultraviolet (UV) radiation. |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the general safety of the test product | Frequency and severity of Adverse Events. |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

#### 1.3 Treatments

| | Test Product | Reference Product |
|---|---|---|
| <b>Product Name</b> | Physiogel Daily Defence<br>Protective Day Cream Light | P3 Standard |
| Product<br>Formulation<br>Code (MFC) | CCI | Commercially Available |
| <b>Expected SPF</b> | 21 | 16 |
| Application Quantity | $2.00 \pm 0.05 \text{ mg} / \text{cm}^2$ | $2.00 \pm 0.05 \text{ mg} / \text{cm}^2$ |
| Route of<br>Administration | Topical | Topical |

### 1.4 Timepoints and visit windows

Deviations from the scheduled assessment times must be avoided. The following are the assessment time windows.

| Visit | Time window |
|---------|--------------------------------------------------------------|
| Visit 2 | 0-7 days after Visit 1 (allowed to be combined with Visit 1) |
| Visit 3 | 1 day after Visit 2 |
| Visit 4 | 0-7 days after Visit 3 (allowed to be combined with Visit 3) |
| Visit 5 | 1 day after Visit 4 |

Visual grading of skin at Visit 3 must happen 16-24 hours after irradiation at Visit 2. Visual grading of skin at Visit 5 must happen 16-24 hours after irradiation at Visit 4.

## 2 Data analysis

Data analysis will be performed by inVentiv Health Clinical. Prior to database hard lock a Blind Data Review Meeting (BDRM) will be conducted in which various aspects of the trial will be discussed and agreed. The statistical analysis software used will be SAS® version 9.4.

All listings will be produced for all randomised subjects, unless otherwise specified.

## 2.1 Populations for analysis

### 2.1.1 Subject disposition

Screen failures will be defined as subjects who consent to participate in the study but are never subsequently randomised. A summary will be provided of the number of subjects screened and the number of screen failures with reasons why subjects were not randomised (Table 14.1.1).



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

Subject disposition will be summarized as the number and percentage of subjects (out of the number of randomised subjects) who complete the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1). The table will also summarize the number and percentage of subjects assigned to each analysis population (refer to section 2.1.3).

#### 2.1.2 Protocol violations

Protocol violations will be tracked by the study team throughout the conduct of the study. All violations will be reviewed prior to un-blinding and closure of the database to ensure all important violations are captured and categorised.

Major violations will be defined in the "Review Listing Requirement (RLR)" document.

A listing of protocol violations will be provided (Listing 16.2.1).

#### 2.1.3 Analysis populations

Five populations are defined below.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | All subjects who are screened | Disposition |
| Subjects | | |
| Randomised | All subjects who are randomised and | Protocol violations |
| | may or may not receive the application of | and data listings |
| | the study products. | |
| Safety | Safety population includes all subjects | Safety analysis |
| | who are randomised and receive any | |
| | application of the study products. | |
| Analysis | The analysis population includes those | SPF analysis |
| Population | randomised subjects who undergo | |
| | irradiation at Visit 4 | |

#### 2.1.4 Subgroups/Stratifications

Not applicable.

#### 2.1.5 Centers pools

Not applicable.

### 2.2 Patient demographics/other baseline characteristics

Demographic and baseline characteristics summaries will be produced for the safety and analysis population.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

#### 2.2.1 Demographic characteristics

Categorical demographic variables include sex, race and Fitzpatrick skin type assessment. These variables will be summarized by the number and percentage of subjects with each relevant characteristic (Table 14.1.2.1 for safety, and Table 14.1.2.3 for analysis population). Age, individual typology angle (ITA°), meanL and meanB values will be summarized by the mean, standard deviation, median, minimum and maximum values. The demographics information age, sex, race, individual typology angle (ITA°), meanL and meanB values will be listed in Listing 16.2.4.1.

The Fitzpatrick scale is a numerical classification that is widely used by dermatologists to classify a person's skin type by their response to the sun exposure.



A tri-stimulus chromameter (Minolta CR 400, Langenhagen, Germany) which utilizes the L\*, a\*, b\* colour space and complies with International Commission on Illumination (CIE) recommendations will be used to measure the colour of each subject's skin (dorsum). Four measurements will be taken on the back of each subject, between the waist and shoulder line, and the individual L\* and b\* values will be recorded as source data. The ITA° will be calculated and recorded on the case report form (CRF) as

calculated and recorded on the case re  
ITA° ={
$$arc\ tangent\ [\frac{(L^*-50)}{b^*}]$$
}  $\frac{180}{3.14159}$ 

#### 2.2.2 General medical history

Medical history data will not be presented in the study report. A data listing will be produced at the blinded data review stage, for evaluation of protocol violations only.

#### 2.2.3 Characteristics of Disease

Not applicable.

<sup>\*</sup>arc tangent is expressed in radians.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | 8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

# 2.3 Treatments (study drug, rescue medication, other concomitant therapies, compliance)

#### 2.3.1 Study Product/drug Compliance and Exposure

Any protocol violations associated with treatment applications will be listed at the blinded data review stage. Any protocol violations leading to exclusion from analysis population will be listed in the Listing 16.2.2.

#### 2.3.2 Concomitant medication

Prior and concomitant medication/non-drug treatments data will be listed in the Listing 16.2.4.2. A data listing will also be produced at the blinded data review stage, for evaluation of protocol violations.

### 2.4 Analysis of Sun Protection Factor (SPF)

#### 2.4.1 Primary efficacy endpoint

#### 2.4.1.1 Primary endpoint definition

The primary analysis will be based on sun protection factor (SPF). Individual SPF for each subject (SPFi) is defined as the ratio of his/her minimal erythemal dose of protected skin (MEDp) over unprotected skin (MEDu), i.e., SPFi = MEDp / MEDu (keeping 1 decimal place for individual SPF). As each subject will have both test product and reference product applied on two sites of dorsum together with an unprotected site, each subject will provide two individual SPFs, one for the test product, one for the reference product. The MEDp at two protected sites and MEDu at the unprotected site of each subject determined by a trained grader at Visit 5 will be used in primary analysis.

Summary statistics for SPF, including mean, standard deviation, will be presented by treatment. The 95% CIs for the mean SPFs of the two treatments will be constructed via t-statistic and presented together with summary statistics (Table 14.2.1.1. for Analysis Population). The study will be considered valid if

- the range of the 95% CI of the mean SPF is within ±17% of the mean SPF for each product;
- The mean SPF of the reference sunscreen formulation (P3) used in the test shall fall within the defined acceptance limits (lower limit, SPF 13.7; upper limit, 17.7).

#### 2.4.1.2 Statistical hypothesis, model, and method of analysis

Except the 95% CI for mean SPF, there is no formal statistical inference to be performed.

#### 2.4.1.3 Supportive analyses

Not applicable.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

#### 2.4.2 Secondary efficacy endpoint

Not applicable.

#### 2.4.3 Handling of missing values/censoring/discontinuations

Missing data will not be replaced or imputed.

#### 2.5 Analysis of secondary objectives

Not applicable.

#### 2.6 Safety

#### 2.6.1.1 Adverse events and Serious Adverse Events

All adverse events (AEs) will be summarised by primary system organ class and preferred term

Treatment emergent adverse events (TEAEs), defined as the AEs reported after study product application, will be summarized by the number and percentage of subjects having any adverse event, any adverse event in each System Organ Class, and and the number of occurrences of each individual adverse event (Table 14.3.1.1). All TEAEs will also be tabulated by severity (Table 14.3.1.2). Treatment emergent AEs suspected of a relationship to study medication will be presented in a similar manner (Table 14.3.1.3). For treatment related AEs, these will also be presented by severity (Table 14.3.1.4).

Deaths occurring during treatment (if any) will be listed (Listing 14.3.2.1) by treatment, including the date and study day of death, and the principal cause of death. Non-fatal serious adverse events causing study treatment discontinuation will be listed (Listing 14.3.2.2).

AEs will be collected from the start of provisional MEDu irradiation procedure until 5 days after the last administration of the study product. SAEs however, if assessed as related to study participation or related to a GSK concomitant medication will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact. All AEs will be listed in Listing 16.2.7.1 for randomised subjects and Listing 16.2.7.2 for non-randomised subjects.

## 2.7 Analysis of other variables

MEDu and MEDp collected from study subjects are used to derive SPF. MEDu and MEDp themselves will not be summarised or analysed. However, a listing for all MED determinations will be provided including the provisional determination (at Visit 3) of the unprotected skin and the final determination (at Visit 5) of both protected and unprotected skin (Listing 16.2.6).



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

## 2.8 Interim analysis

There is no formal interim analysis. The procedure described in sample size determination will be performed by site staff.

### 2.9 Sample size calculation

Healthy volunteers aged between 18-70 years (inclusive) with Fitzpatrick phototype I, II or III, an ITA° value greater than 28° and who are untanned on the test area will be recruited for this study. The study will contain a population of subjects of more than one Fitzpatrick phototype.

To complete the study successfully, the minimum number of valid individual sun protection factor (SPFi) results will be 10 and the maximum number of valid SPFi results will be 20 for both the test product and positive control. In order to achieve between 10 and 20 valid SPFi results, a maximum of 5 individual invalid results may be excluded from the calculation of the mean SPF. Consequently, the actual number of subjects used for the study will fall between a minimum of 10 and a maximum of 25 (i.e. a maximum of 20 valid SPFi results plus 5 rejected invalid results).

In order to determine the number of test subjects, the 95% confidence interval (95% CI) of the mean SPF shall be taken into account. A minimum of 10 subjects shall be tested. The test shall be considered valid for the first 10 subjects if the resulting range of the 95% CI of the mean SPF is within  $\pm 17\%$  of the mean SPF. If it is not within  $\pm 17\%$  of the mean SPF, the number of subjects shall be increased stepwise from the minimum number of 10 until the 95% CI statistical criterion is met (up to a maximum of 20 valid results from a maximum of 25 subjects tested). If the statistical criterion has not been met after 20 valid results from a maximum of 25 subjects, then the test shall be rejected.

## 3 Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol version 1.0 [(Dated: 28/Mar/2017)].



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

# 4 Appendix 1:

# 4.1 List of Tables, Listings and Figures

## 4.2 Tables

| Table Number | Table Title (Population) | Template |
|---|---|---|
| 14.1.1 | Subject Disposition (All Screened Subjects) | Appendix 2 |
| 14.1.2.1 | Subject Demographics and Baseline Characteristics | Appendix 2 |
| | (Safety Population) | |
| 14.1.2.2 | Subject Demographics and Baseline Characteristics | 14.1.2.1 |
| | (Analysis Population) | |
| 14.2.1.1 | Summary of Sun Protection Factor by Treatment | Appendix 2 |
| | (Analysis Population) | |
| 14.3.1.1 | Treatment Emergent Adverse Events (Safety | Appendix 2 |
| | Population) | |
| 14.3.1.2 | Treatment Emergent Adverse Events by Severity | Appendix 2 |
| | (Safety Population) | |
| 14.3.1.3 | Treatment Emergent Treatment Related Adverse | 14.3.1.1 |
| | Events (Safety Population) | |
| 14.3.1.4 | Treatment Emergent Treatment Related Adverse | 14.3.1.2 |
| | Events by Severity (Safety Population) | |

4.3 Listings

| Listing Number | Listing Title (Population) | Template |
|----------------|-----------------------------------------------|------------|
| 14.3.2.1 | Listing of Deaths (Randomised population) | 16.2.7.1 |
| 14.3.2.2 | Listing of Serious Adverse Events leading to | 16.2.7.1 |
| | Discontinuation (Randomised population) | |
| 16.1.7 | Randomisation Information (Randomised | Appendix 2 |
| | Population) | |
| 16.2.1 | Individual Subjects Protocol Violations | Appendix 2 |
| | (Randomised Population) | |
| 16.2.2 | Protocol Violations Leading to Exclusion from | Appendix 2 |
| | Analysis Population (Randomised Population) | |
| 16.2.4.1 | Demographic Characteristics | Appendix 2 |
| | (Randomised Population) | |
| 16.2.4.2 | Prior and Concomitant Medications | Appendix 2 |
| | (Randomised Population) | |
| 16.2.4.3 | Listing of the identification for Technician | Appendix 2 |
| | (Randomised Population) | |
| 16.2.6 | Individual Subject Efficacy Data (Randomised | Appendix 2 |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Statistical Analysis Plan Forte/207640

| <b>Listing Number</b> | Listing Title (Population) | Template |
|---|---|---|
| | Population) | |
| 16.2.7.1 | All Adverse Events (Randomised Population) | Appendix 2 |
| 16.2.7.2 | All Adverse Events (Non-Randomised Subjects) | 16.2.7.1 |

Note: If there are no data to display generate a null listing.

# 4.4 Top line Outputs:

| Table/Listing | Table/Listing/Figure Title (Population) |
|---|---|
| Figure Number | |
| 14.1.1 | Subject Disposition (All Screened Subjects) |
| 14.1.2.1 | Subject Demographics and Baseline Characteristics (Safety Population) |
| 14.2.1.1 | Summary of Sun Protection Factor by Treatment (Analysis Population) |
| 14.3.1.1 | Treatment Emergent Adverse Events (Safety Population) |
| 16.2.7.1 | All Adverse Events (Randomised Population) |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 11: | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | |


# 5 Appendix 2:

## 5.1 Templates for the Tables, Listings and Figures

This is a guideline which will give the guidance of treatment labels that will be used for the table header and in the figures, listings and in the footnotes.

The treatment labels for the column headings will be as follows:

- Physiogel Daily Defence
- P3 Standard



| Document Name | 16.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | |


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

Table 14.1.1 Subject Disposition All Screened Subjects

| A <u>ll</u> Screened Subjects (N=XX) | |
|--------------------------------------|---------------|
| | Overall(N=XX) |
| | n (%) |
| TOTAL NUMBER OF SUBJECTS SCREENED | xx |
| SUBJECTS NOT RANDOMISED | Xx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xx (xx.x) |
| ADVERSE EVENTS | xx (xx.x) |
| LOST TO FOLLOW UP | xx (xx.x) |
| PROTOCOL DEVIATION | xx (xx.x) |
| WITHDRAWAL OF CONSENT | xx (xx.x) |
| OTHER | xx (xx.x) |
| SUBJECTS RANDOMISED | xx (xx.x) |
| COMPLETED | xx (xx.x) |
| DID NOT COMPLETE | xx (xx.x) |
| DID NOT MEET STUDY CRITERIA | |
| ADVERSE EVENT | xx (xx.x) |
| LOST TO FOLLOW UP | xx (xx.x) |
| PROTOCOL DEVIATION | xx (xx.x) |
| WITHDRAWAL OF CONSENT | xx (xx.x) |
| OTHER | xx (xx.x) |



| Document Name | 16.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 11:01: | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | |

Confidential Page 17

Forte/207640

| | Overall(N=XX) |
|--------------------|---------------|
| | n (%) |
| DOMISED POPULATION | xx (xx.x) |
| TY POPULATION | xx (xx.x) |
| LYSIS POPULATION | xx (xx.x) |

Program: PPD Source: PPD

For Non-Randomised section percentages has been calculated based on total number of subjects screened. For Randomised section percentages has been calculated based on total number of subjects randomised.

Note to programmer: For subjects not randomised and subjects not completing the study, the reasons should be consistent with the reasons in eCRF.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 11:0 | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | |


Forte/207640


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

# Table 14.1.2.1 Subject Demographics and Baseline Characteristics Safety Population

| Safety Population (N=XX) | |
|-------------------------------------------|-----------------|
| | Overall Overall |
| | (N=XX) |
| SEX n (%) | |
| MALE | xx (xx.x) |
| FEMALE | xx (xx.x) |
| RACE n (%) | |
| ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | xx (xx.x) |
| AFRICAN AMERICAN/AFRICAN HERITAGE | xx (xx.x) |
| AMERICAN INDIAN OR ALASKAN NATIVE | xx (xx.x) |
| NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x) |
| WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | xx (xx.x) |
| (include all captured as in eCRF) | xx (xx.x) |
| AGE (YEARS) | |
| n | XX |
| MEAN | XX.X |
| SD | XX.XX |
| MEDIAN | XX.X |
| MINIMUM | XX |



| Document Name | 6.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 11:01:02 | |
| Reason For Issue | Imported as Effective from Legacy System | |
| Confidential | Page 1 | 9 |

Forte/207640

| | Overall Overall |
|------------------------------------------|-----------------|
| | (N=XX) |
| MAXIMUM | XX |
| TEXTION | |
| ITAº | VV |
| n | XX |
| MEAN | XX.X |
| SD | XX.XX |
| | XX.X |
| MEDIAN | XX |
| MINIMUM | |
| MAXIMUM | XX |
| FITZPATRICK SCALE FOR SKIN TYPE | |
| I = ALWAYS BURNS EASILY: NEVER TANS | xx (xx.x) |
| II = ALWAYS BURNS EASILY: TANS MINIMALLY | xx (xx.x) |
| III = BURNS MODERATELY: TANS GRADUALLY | xx (xx.x) |
| IV = BURNS MINIMALLY: ALWAYS TANS WELL | xx (xx.x) |
| V = RARELY BURNS: TANS PROFUSELY | xx (xx.x) |
| VI = NEVER BURNS: DEEPLY PIGMENTED | xx (xx.x) |

Program: PPD Source: PPD

Programming Note: The similar descriptive statistics should be provided for meanL\* and meanb\*.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | |
|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective 090032d580dcf91b (8-Dec-2017 11 | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | |


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

# Table 14.2.1.1 Summary of Sun Protection Factor by Treatment Analysis Population

| A <u>nalysis</u> | Population | (N=XX) |
|------------------|------------|--------|
| | - | |

| Visit | Variable | Physiogel Daily Defence | P3 Standard |
|---|---|---|---|
| | | (N=XX) | (N=XX) |
| VISIT 5 | n (number of invalid<br>cases) | xx | XX |
| | | Summary for Valid Case | s |
| | n (number of valid cases) | xx | xx |
| | MEAN | x.xx | x.xx |
| | SD | x.xxx | x.xxx |
| | 95% CI | (x.xx, x.xx) | (x.xx, x.xx) |
| | CI[%] | XX.X | xx.x |

Program: PPD Source: PPD

Note to programmer: 1. Keep two decimal places for mean, 95% CI.

2. Keep three decimal places for SD.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

Table 14.3.1.1
Summary of Treatment Emergent Adverse Events
Safety Population

| Safety Population (N=xx) | | Sureey 1 opt | 414(10) | | |
|---|---|---|---|---|---|
| System Organ Class and<br>Preferred Term | Physiogel Daily Defence (N=XX) | | P3 Standard | Overall (N=XX) | |
| | | | (N=XX) | | |
| <del>-</del> | n (%) | nAE | | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT<br>LEAST ONE AE | xx (xx.x) | xx | ••• | xx (xx.x) | xx |
| NUMBER OF SUBJECTS WITH NO AE | xx (xx.x) | XX | | xx (xx.x) | xx |
| SKIN AND SUBCUTANEOUS TISSUE DISORDERS | xx (xx.x) | xx | | xx (xx.x) | xx |
| ERYTHEMA | xx (xx.x) | xx | ••• | xx (xx.x) | XX |
| DERMATITIS | xx (xx.x) | XX | ••• | xx (xx.x) | xx |
| GASTROINTESTINAL SYSTEM | xx (xx.x) | XX | ••• | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | xx | ••• | xx (xx.x) | xx |
| DRY MOUTH | xx (xx.x) | xx | ••• | xx (xx.x) | XX |
| VOMITING | xx (xx.x) | xx | | xx (xx.x) | XX |

n (%) = Number (percent) of subjects; nAE = Number of adverse events.

Program: PPD Source: PPD



| Document Name | cument Name 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | 8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Safety Population (N=xx)

Protocol: 207640

Page x of y
Program Run Date:ddmonyyyy

Table 14.3.1.2 Summary of Treatment Emergent Adverse Events by Severity Safety Population

| System Organ Class and<br>Preferred Term | | Р | hysiogel Dai | ly Defen | ice | | P3 Standard | | | | Overall | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=X) | () | | | (N=XX) | | | | (N=XX) | | |
| | Mild | | Moderat | te | Seve | re | | Milo | d | Moder | rate | Seve | re |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE | | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE<br>AE | xx (xx.x) | XX | xx (xx.x) | xx | xx<br>(xx.x) | xx | ••• | xx<br>(xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| | | XX | | XX | | XX | • • • | | XX | | XX | | XX |
| SKIN AND SUBCUTANEOUS TISSUE<br>DISORDERS | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | | xx<br>(xx.x) | xx | xx<br>(xx.x) | XX | xx (xx.x) | xx |
| ERYTHEMA | xx (xx.x) | XX | xx (xx.x) | XX | xx<br>(xx.x) | XX | ••• | xx<br>(xx.x) | XX | xx<br>(xx.x) | XX | xx (xx.x) | XX |
| DERMATITIS | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | ••• | xx<br>(xx.x) | XX | (xx.x) | xx | xx (xx.x) | xx |
| GASTROINTESTINAL SYSTEM | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | ••• | xx<br>(xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| ABDOMINAL PAIN | xx (xx.x) | xx | xx (xx.x) | xx | xx<br>(xx.x) | xx | ••• | xx<br>(xx.x) | xx | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| DRY MOUTH | xx (xx.x) | xx | xx (xx.x) | XX | xx<br>(xx.x) | XX | ••• | xx<br>(xx.x) | XX | xx<br>(xx.x) | xx | xx (xx.x) | xx |
| VOMITING | xx (xx.x) | XX | xx (xx.x) | XX | xx<br>(xx.x) | xx | ••• | xx<br>(xx.x) | xx | `xx (<br>(xx.x) | xx | xx (xx.x) | xx |

n (%) = Number (percent) of subjects; nAE = Number of adverse events.

Program: PPD Source: PPD



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| Туре | Version | <b>Document Identifier</b> | Effective Date |
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | 8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Forte/207640


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

Listing 16.1.7
Randomisation Information
Randomised Population

| Subject | Age/Sex/Race[1] | Randomisation Number | Test Site/Treatment | Date of randomisation (dd/mmm/yyyy) |
|---|---|---|---|---|
| Number | | | Randomised | |
| PPD | | | | PPD |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

Program: PPD Source: PPD

Note to programmer: Check actual races captured in eCRF to adjust the race name and abbreviations



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |

Confidential Page 24

Forte/207640

Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

# Listing 16.2.1 Individual Subjects Protocol Violations Randomised Population

| Subject<br>Number | Age/Sex/Race[1] | Visit | Deviation Sequence | Protocol Deviation |
|---|---|---|---|---|
| PPD | | 3 | 1 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Program: PPD Source: PPD

Note to programmer: Check actual races captured in eCRF to adjust the race name and abbreviations

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| Туре | Version | <b>Document Identifier</b> | Effective Date |
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

Listing 16.2.2

# $\begin{array}{c} {\tt Protocol\ Violations\ Leading\ to\ Exclusion\ from\ Analysis\ Population} \\ {\tt Randomised\ Population} \end{array}$

| Subject<br>Number | Deviation<br>Sequence | Start Date | End Date | Deviation Description |
|---|---|---|---|---|
| PPD | 1 | 28MAR2017 | 28MAR2017 | XXXXXXXX |

Program: PPD Source: PPD



| Document Name 16.1.7 Documentation of statistical methods.pdf | | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

Listing 16.2.4.1

Demographic Characteristics Randomised Population

| Subject Number | Age | Sex | Race | MeanL* | Meanb <sup>*</sup> | ITA <sup>0</sup> Value | FITZPATRICK SCALE FOR SKIN TYPE |
|---|---|---|---|---|---|---|---|
| PPD | | | | 69.03 | 55.1 | 55.7 | I = ALWAYS BURNS EASILY: |
| | | | | | | | NEVER TANS |

•••••••

Program: PPD Source: PPD



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |
| Confidential | Page 2 | 7 | |

Forte/207640

Protocol: 207640

Page x of y
Program Run Date:ddmonyyyy

Listing 16.2.4.2

Prior and Concomitant Medications Randomised Population

| Subject<br>Number | Screening<br>Date | Medication | Dosage | Reason for<br>Medication | Medication<br>Start<br>Date [1] | Medication<br>End<br>Date [1] | Ongoing<br>Status<br>Yes/No |
|---|---|---|---|---|---|---|---|
| PPD | | | 10MG PO OD | HIGH BLOOD<br>PRESSURE | 2011 | CONTINUING | YES |

[1] Only known parts of partial dates are listed.

Program: PPD Source: PPD



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Forte/207640


Protocol: 207640

Page x of y
Program Run Date:ddmonyyyy

Listing 16.2.4.3

Listing of the Identification for Technician Randomised Population

| Subject Number | Irradiation at Visit 2 | Visual Grading at Visit 3 | Product Application and Irradiation at Visit 4 | Visual Grading at Visit 5 |
|---|---|---|---|---|
| PPD | AP | AP | AP | AP |

Program: PPD Source: PPD

Programming Note: The AP is just an example, please use the real data while creating the listing.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | (8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Forte/207640


Protocol: 207640

Page x of y Program Run Date:ddmonyyyy

#### Listing 16.2.6 Individual Subjects Efficacy Data Randomised Population

| Subject | Age/Sex/Race[1] | Visit | Test- | Sub-Site | Treatment | Variable | Variable Value | Valid / | Exclusion Justification |
|---|---|---|---|---|---|---|---|---|---|
| Number | | | Site | | | | | Excluded | |
| PPD | | | | | | Provisional | x.xx | | |
| | | | | | | MEDu | | | |
| | | | | | | MEDu | x.xx | | |
| | | | | | | MEDp test | x.xx | | |
| | | | | | | MEDp reference | x.xx | | |
| | | | | | | SPFi test | XX.X | Valid | |
| | | | | | | SPFi reference | XX.X | excluded | invald fortest product |
| | | | | | | Provisional | x.xx | | |
| | | | | | | MEDu | | | |
| | | | | | | MEDu | x.xx | | |
| | | | | | | MEDp test | x.xx | | |
| | | | | | | MEDp reference | x.xx | | |
| • • • | | | | | | SPFi test | XX.X | | |
| | | | | | | SPFi reference | XX.X | | |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

Program: PPD Source: PPD

Note to programmer: Check actual races captured in eCRF to adjust the race name and abbreviations.



| Document Name | 16.1.7 Documentation of statistical methods.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91b | 8-Dec-2017 11:01:02 |
| Reason For Issue | Imported as Effective from Legacy System | | |


Forte/207640


Protocol: 207640

Page x of v Program Run Date:ddmonvvvv

Listing 16.2.7.1 All Adverse Events Randomised Population

Treatment Group: Physiogel Daily Defence/no treatment

| Subject<br>Number | Age/Sex/R<br>ace[1] | Adverse Event (Preferred Term) (System Organ Class) | Start Date<br>/Study<br>Day[2] | Start Time | End<br>Date | End<br>Time | Frequency<br>/Intensity<br>[3] | Related to<br>Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcom<br>e | Serious<br>? | Withdrew?[<br>4] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | | | PPD | | | Singl<br>e/<br>MILD | No | NOT<br>APPLICAB<br>LE | RECOVE<br>RED/RE<br>SOLVED | NO | NO |

[1] Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

- [2] Study day is the day relative to start of treatment, day 1 being the day of first treatment.
- [3] INT = Intermittent and SGLE = Single.
- [4] Did subject withdraw from study as a result of this adverse event?

Source: ppn Program: ppp

Programming Note: Those AEs are not coming under treatment, that will displayed under the overall treatment group.

Programming Note for Listing 16.2.7.2:

- ☐ Repeat the same layout for listing 16.2.7.2
- Population should be used 'Non randomised Subjects'
- The fourth column should be only 'Start Date'
- Delete the footnote related to study day and adjust the numbers accordingly.



| Document Name | 16.1.71 SAP Signatures.pdf | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580dcf91a | (8-Dec-2017 11:00:52 |
| Reason For Issue | Imported as Effective from Legacy System | | |

| inVentiv | Client Approval Form: Final Statistical Analysis |
|----------|--------------------------------------------------|
| Health | Plan Shells |

| | Project Identifiers |
|------------------------|--------------------------------------------|
| Client: GSKCH | Protocol No.: 207640 |
| Project ID Code: PPD | Protocol Version (date): 1.0 (28-MAR-2017) |
| SAP Version: 1.0 | SAP Author: PPD |
| SAP Date : 29-JUN-2017 | |

The signatures below acknowledge that the Statistical Analysis Plan Shells prepared by inVentiv Health for GSKCH are final.



Confidential 1 of 1